CLINICAL TRIAL: NCT02611765
Title: Syphilis Response to Higher Penicillin Dosage in HIV Co-Infected Patients
Brief Title: Syphilis Response to Higher Penicillin Dosage: The 2.4 Versus 7.2 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jose Serpa-Alvarez, Co-Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22816
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced therapy (Experimental): Benzathine penicillin G intramuscular 7.2 million units Three doses of 2.4 million units of intramuscular benzathine penicillin G administered weekly (a total of 7.2 million units)
  Interventions: Drug: Benzathine penicillin G intramuscular 7.2 million units
- Standard therapy (Active Comparator): Benzathine penicillin G intramuscular 2.4 million units A single intramuscular injection of 2.4 million units of benzathine penicillin G
  Interventions: Drug: Benzathine penicillin G intramuscular 2.4 million units

INTERVENTIONS:
Drug: Benzathine penicillin G intramuscular 7.2 million units — Three doses of intramuscular 2.4 million units of benzathine penicillin G administered weekly (a total of 7.2 million units).
  Other Names: Enhanced therapy
  Arms: Enhanced therapy
Drug: Benzathine penicillin G intramuscular 2.4 million units — A single dose of intramuscular 2.4 million units of benzathine penicillin G
  Other Names: Standard therapy
  Arms: Standard therapy

SUMMARY:
Syphilis remains a significant health problem worldwide, with an estimated 10.6 million new cases per year. Due to shared transmission route and risk factors, co-infection with syphilis and Human Immunodeficiency Virus (HIV) is not uncommon. Several studies have evaluated the response to syphilis treatment in HIV-infected patients. They support the claim that patients with HIV have a slower decrease in syphilis antibody titers, and that they may progress to neurosyphilis in earlier stages.

The Center for Disease Control and Prevention's Sexually Transmitted Disease Treatment Guidelines has advocated treating HIV-infected patients who have primary, secondary syphilis or early latent syphilis with the same doses of penicillin as for HIV-uninfected patients (single dose of 2.4 million units of benzathine penicillin G). The investigators designed a randomized controlled trial in order to compare the efficacy of three- versus single-dosed regimens of intramuscular benzathine penicillin G (BPG) for the treatment of early syphilis in HIV-infected patients.

DETAILED DESCRIPTION:
The investigators conducted a prospective, randomized, open label study at three clinical sites including Thomas Street Health Center and North West Clinic (Harris Health System), and the Michael E. DeBakey Veterans Affairs Medical Center in Houston, Texas. After obtaining written informed consent, the investigators randomly assigned patients to either a single intramuscular injection of 2.4 million units of BPG (standard therapy) or three doses (enhanced therapy) of intramuscular BPG administered weekly (a total of 7.2 million units).

Patients were eligible for inclusion in the study if they were 18 years of age or older and had a diagnosis of HIV. The diagnosis of syphilis was made based on a positive Rapid Plasma Reagin (RPR) and treponema pallidum particle agglutination tests. Patients with primary, secondary and early latent syphilis were included.

Exclusion criteria were history of penicillin allergy, diagnosis of late latent syphilis, neurosyphilis, and antibiotic use with significant activity against Treponema pallidum within the preceding two weeks.

Follow-up period was 12 months. Serum samples were obtained at initial visit and follow-up visits every 3 months for serological testing for syphilis. Treatment success was defined as a decrease in RPR titer of >= 2 dilutions (4-fold) from the initial RPR titer during the follow-up period.

Both intention-to-treat and per-protocol analyses were performed

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV by ELISA and confirmed by Western blot
* Positive Rapid Plasma Reagin and treponema pallidum particle agglutination tests

Exclusion Criteria:

* History of penicillin allergy
* Diagnosis of late latent syphilis
* Diagnosis of neurosyphilis
* Antibiotic use with significant activity against Treponema pallidum within the preceding two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Serpa-Alvarez, MD, Principal Investigator — Assistant Professor (Medicine: Infectious Disease)

REFERENCES:
- [Derived] Andrade R, Rodriguez-Barradas MC, Yasukawa K, Villarreal E, Ross M, Serpa JA. Single Dose Versus 3 Doses of Intramuscular Benzathine Penicillin for Early Syphilis in HIV: A Randomized Clinical Trial. Clin Infect Dis. 2017 Mar 15;64(6):759-764. doi: 10.1093/cid/ciw862. PMID 28200045

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Therapy: Three doses of 2.4 million units of intramuscular benzathine penicillin G administered weekly (a total of 7.2 million units)
  Enhanced therapy: Three doses of intramuscular 2.4 million units of benzathine penicillin G administered weekly (a total of 7.2 million units).
- Standard Therapy: A single intramuscular injection of 2.4 million units of benzathine penicillin G
  Standard therapy: A single dose of intramuscular 2.4 million units of benzathine penicillin G
Period: Overall Study
Arm/Group | Enhanced Therapy | Standard Therapy
Started | 29 | 35
Completed | 27 | 29
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Therapy | Standard Therapy | Total
Number analyzed (Participants) | 29 | 35 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11) | 35 (10) | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 27 | 34 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  Whites | 1 | 6 | 7
  African Americans | 15 | 22 | 37
  Hispanics | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Defined as a Decrease in Rapid Plasma Reagin (RPR) Titer of >= 2 Dilutions (4-fold)
Description: Number of participants who achieve treatment success. Loss to follow-up was assumed to be a failure.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Enhanced Therapy | Standard Therapy
Number analyzed (Participants) | 29 | 35
participants | 27 | 28

ADVERSE EVENTS:
Arm/Group | Enhanced Therapy | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No